CLINICAL TRIAL: NCT01441375
Title: Complications in Patients With Sickle Cell Disease and Utilization of Iron Chelation Therapy: A Retrospective Medical Records Review
Brief Title: Sickle Cell Disease: A Retrospective Chart Review
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CICL670A2418
Record Dates: First submitted 2011-09-07; First posted 2011-09-27 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Sickle Cell Anemia
Keywords: Sickle cell anemia
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Sickle cell patients non-transfused
- Sickle cell patients transfused with no ICT
- Sickle cell patients transfused with ICT

SUMMARY:
This study is a retrospective chart review of sickle cell patients and will include patients whom have received blood transfusions and those whom have not. Of the transfused patients, it will also include those whom have received chelation therapy and those whom have not.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of Sickle Cell Disease (SCD) and a confirmed genotype
2. Patients ≥ 16 years of age
3. Patients with ≥ 6 months of follow-up data available from first SCD treatment at the center after they reach 16 years old
4. At least one SF reading during a non-acute phase on or after the first SCD treatment at the center after they reach 16 years old

Exclusion Criteria:

1. Patients who participated in a clinical trial for an iron chelating medication or in a clinical trial for transfusions for SCD (1) within the six months before the index date or (2) during the patient observation period
2. Patients with sickle cell trait

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Sickle cell anemia
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Sickle cell complications | average of 5 years

SECONDARY OUTCOMES:
Utilization of health care delivery to treat sickle cell complications | average of 5 years
Overall survival | average of 5 years
Utilization of blood transfusions (patients with frequent transfusions only) | average of 5 years
Burden of iron overload (patients with frequent transfusions only) | average of 5 years
Utilization of Iron Chelation Therapies (ICTs) (patients receiving deferoxamine or deferasirox [Exjade®] only) | average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Tulane University, New Orleans, Louisiana
  - Universit of Tennessee, Memphis, Tennessee